CLINICAL TRIAL: NCT03135925
Title: Is it Feasible to Conduct a Randomised Controlled Trial of Pre Transplant Exercise (Pre-habilitation) for Multiple Myeloma Patients Awaiting Autologous Stem Cell Transplantation?
Brief Title: Feasibility of Pre Transplant Exercise (Pre-habilitation) for Multiple Myeloma Patients Awaiting Autologous Stem Cell Transplantation
Acronym: PREeMPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STH18154
Record Dates: First submitted 2016-09-27; First posted 2017-05-02 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Myeloma
MeSH Terms: conditions — Neoplasms, Plasma Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Other): Exercise program
  Interventions: Other: Supervised Exercise Program

INTERVENTIONS:
Other: Supervised Exercise Program — Participants will be invited to attend a weekly supervised exercise program over six weeks, in the time before their bone marrow transplantation

SUMMARY:
The investigators propose to determine whether it is acceptable to patients with a diagnosis of multiple myeloma (a type of blood cancer that can cause bone weakness, pain and fatigue) to be offered and attend an exercise group before receiving an autologous stem cell transplantation (being given back one's own stem cells, following receipt of intensive chemotherapy, to enable bone marrow to start producing blood cells again). Exercise has been shown to be effective in reducing many of the side effects of myeloma and the treatment patients receive to manage the disease. Prehabilitation i.e. providing an intervention after diagnosis but before treatment begins has been effective in reducing the severity of side effects of treatment in cancer patients receiving surgery. No evidence exists for its use in patients with myeloma. Patients awaiting transplantation will be provided with information regarding the study and invited to join. Patients who agree to take part will attend the hospital for an assessment of their exercise capability and to complete one set of four questionnaires. They will receive an exercise booklet, advice and complete one attempt at their exercise programme under supervision of a physiotherapist. Patients will be requested to attend the gym for a minimum of six further weeks to complete their exercise programme. Patients will complete a repeat set of questionnaires and a repeat walking test six weeks after the first, on admission to hospital for their transplant and on the day they leave hospital. Some patients will be invited to discuss their opinions of the exercise programme and how useful they felt it was to them in preparing for their transplant. If the study shows that the exercise programme is acceptable to patients and we can recruit enough patients to test it in a larger trial, the investigators will apply for further funding.

ELIGIBILITY:
Inclusion Criteria:

* All patients will have a diagnosis of multiple myeloma and assigned to the autologous transplantation waiting list for either a first or second transplant

Exclusion Criteria:

* History of unstable angina or a heart attack in the previous month to allow safe completion of the six minute walk test.
* Medical stability is a pre-requisite for transplantation so no patients would be excluded on this basis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of exercise sessions attended | 12 months
  this is a feasibility study, so monitoring attendance at the study will be the primary outcome measure

SECONDARY OUTCOMES:
Six minute walking distance | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  Six minute walking distance
Mental well-being | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  Warwick and Edinburgh Mental Well-being Scale
Physical Activity/fitness 1 | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  Godin Leisure Time
Physical Activity/fitness 2 | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  International Physical Activity Questionnaire
Quality of Life 1 | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  FACT-MM
Quality of Life 2 | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  EORTC QLQ C30 MY20
Self-efficacy with exercise | At initial assessments and 6th and final exercise session, which will be between 6 and 12 weeks from initial assessment
  SCI Self Efficacy for Exercise Scale

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mawson, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keen C, Skilbeck J, Ross H, Smith L, Collins K, Dixey J, Walters S, Greenfield DM, Snowden JA, Mawson S. Is it feasible to conduct a randomised controlled trial of pretransplant exercise (prehabilitation) for patients with multiple myeloma awaiting autologous haematopoietic stem cell transplantation? Protocol for the PREeMPT study. BMJ Open. 2018 Mar 9;8(3):e021333. doi: 10.1136/bmjopen-2017-021333. PMID 29525775
- [Derived] Mawson S, Keen C, Skilbeck J, Ross H, Smith L, Dixey J, Walters SJ, Simpson R, Greenfield DM, Snowden JA. Feasibility and benefits of a structured prehabilitation programme prior to autologous stem cell transplantation (ASCT) in patients with myeloma; a prospective feasibility study. Physiotherapy. 2021 Dec;113:88-99. doi: 10.1016/j.physio.2021.08.001. Epub 2021 Aug 5. PMID 34563917